CLINICAL TRIAL: NCT06018220
Title: Percutaneous Dilatational Tracheostomy vs. Surgical Tracheostomy in Neurocritically Ill Patients - a Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Birgitte Majholm, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: NEU6021
Record Dates: First submitted 2023-08-11; First posted 2023-08-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Tracheostomy Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present quality study is to examine the relationship between choice of tracheotomy procedure and complications in a neurocritically ill patient population at a single center. Secondary outcomes are the influence of clinician skill level (for PDTs), time from admission to tracheostomy, length of stay and time to decannulation.

DETAILED DESCRIPTION:
Neurocritically ill patients often require placement of a tracheostomy at some point during admission, as impaired consciousness and insufficient protective airway reflexes often make weaning from mechanical ventilation prolonged.

Percutaneous dilatational tracheostomy (PDT) with fiberoptic visualization can be performed bedside by neurointensivists or residents under supervision, unless there are contraindications. However, concerns regarding tracheal stenosis following PDT have been raised. This a rare complication but when it occurs it is a severe long-term complication, and the patients are often in need of repeated interventions. The alternative is surgical tracheostomy (ST) which is more resource intensive but perceived as safer in high risk patients. The indication for tracheostomy (and the choice of procedure) is ultimately based on judgement of clinical team.

Systematic reviews have found no difference between PDT and ST regarding severe complications, apart from a higher incidence of wound infections after ST. However, a higher incidence of complications following PDT has been reported when residents are performing the procedure, suggesting an influence of physician skill level.

Methods:

This is a retrospective observational single-center quality study. All patients > 18 years of age admitted to the Neurointensive Care Unit at Rigshospitalet, Copenhagen between January 2018 and December 2022 with a registered procedure code for either PDT or ST wil be included. Approval from departmental leadership and The Judicial Department at Rigshopitalet has been attained. Data will be extracted from the electronical medical records and any short (< 1 week) or long-term complications will be registered. The follow-up period is 6 months.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to Neurointensive Care Unit, Rigshospitalet, Denmark AND having a tracheostomy performed during their stay.

-

Exclusion Criteria:

Children - age < 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patientiens in Neurointensive Care. Diagnosis are: Traumatic brain injury, intracranial haemorrhage, subarachoid haemorrahge, spinal cord injury, guillian barre, myastenia gravis, status epilepticus, postoperative conditions.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complications following tracheostomy | Up to 1 week after tracheostomy procedure
  Bleeding; pneumothorax, pneumomediastinum, lost airway, via falsa, procedure-related death, other.
Number of patients with complications following tracheostomy - long term. | From 1 week up to 6 months after the tracheostomy procedure
  Tracheal stenosis, fistula, wound infection, accidental decannulation, scarring, delayed wound healing, changes in voice or speech, other.

SECONDARY OUTCOMES:
Number of complications according to the skilled level of the clinician performing the tracheostomy (only for percutaneous dilatational tracheostomy) | Up to 6 months following tracheostomy
  Non-skilled residents vs. senior physician
Days | Up to 6 months
  Time from admission to tracheostomy, time to decannulation, time to discharge from ICU/hospital

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Soerensen, PHD, Study Chair — Department of Neruoanaesthesiology
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No